CLINICAL TRIAL: NCT01094002
Title: Effects of a Structured Occupational Therapy Intervention in an Acute Geriatric Unit. A Randomised Clinical Trial
Brief Title: Effects of a Structured Occupational Therapy Intervention in an Acute Geriatric Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Collaborators: Instituto Ciencias de la Salud, Junta de Comunidades de Castilla-La Mancha (Unknown)
Responsible Party: Pedro Abizanda Soler, Complejo Hospitalario Universitario de Albacete
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI02069-00
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-02

CONDITIONS: Occupational Therapy
Keywords: OCCUPATIONAL THERAPY; RANDOMISED CLINICAL TRIAL; AGED; PATIENT CARE

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occupational therapy intervention (OTI) (Experimental): 198 subjects. The OTI schedule consisted of a daily 45-minute session, Monday through Friday, for the duration of hospitalisation. Activities were carried out in a structured manner and varied according to need and day of admission. On the first day, the patient's needs were analysed, including the need for iatrogenic prevention, retraining in basic and instrumental activities of daily living, technical aids, instruct the primary caregiver in patient mobilisation techniques, and social and occupational motivation. All OTI participants received an average of 5 sessions during hospitalisation.
  Interventions: Other: Occupational therapy intervention
- Conventional treatment model group (No Intervention): 202 subjects. All subjects received medical treatment, nursing care, physical therapy, and social assistance in accordance with the usual practice of the geriatrics unit.

INTERVENTIONS:
Other: Occupational therapy intervention — Day 1: Physical, functional, cognitive, social, and emotional assessment. Need analysis for iatrogenic prevention, retraining in BADL and IADL, technical aids, instructions in patient mobilisation techniques, and for social and occupational motivation.
  Day 2 until discharge: 45-minute sessions. Cognitive stimulation and confusional syndrome prevention, instructions to the caregivers on how to prevent complications such as immobility, delirium, falls, urinary incontinence, or pressure sores, and patient stimulation, retraining in activities of daily living.
  Day of discharge: Instruction for caregivers on managing the patient's residual deficits, assessment for technical aids, recommendations for patient increased independence in ADL, and social and occupational activities.
  Arms: Occupational therapy intervention (OTI)

SUMMARY:
Objectives: To compare the benefits of structured occupational therapy intervention by a single geriatric therapist with the benefits of the conventional treatment model in the functional recovery of patients admitted to an acute geriatric unit.

Design: Non-pharmacological randomised clinical trial. Setting: Acute Geriatric Unit, Albacete, Spain. Participants: The trial included 400 patients admitted consecutively over 6 months to an acute geriatric unit for acute illness or exacerbation of a chronic medical condition. Participants were randomised to the occupational therapy intervention or conventional treatment model group; 198 patients received occupational therapy. All patients completed the study. The mean age was 83.5, and 56.8% were women.

Interventions: Needs assessment, iatrogenic prevention, retraining in basic and instrumental activities of daily living, assessment of need for technical aids, instruction for primary caregiver in patient mobilisation techniques, and structured social and occupational motivation as per protocol in three groups of patients (cardiopulmonary disease, stroke, and other conditions) 5 days a week, 30 to 45 minutes a day over the entire hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 65 or older consecutively admitted to the acute geriatric unit at the Complejo Hospitalario Universitario in Albacete, Spain, between November 2002 and June 2003 for an acute medical illness or exacerbation of a previous chronic condition

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Functional recovery | The day of discharge from hospitalization (average 10 days)
  Recovery of 10 or more Barthel index points

SECONDARY OUTCOMES:
Confusional status | The day of discharge from hospitalization (average 10 days)
  Confusion Assessment Method
Death | The day of discharge from hospitalization (average 10 days)
Hospital stay | The day of discharge from hospitalization (average 10 days)
Upper limb function improvement | The day of discharge from hospitalization (average 10 days)
  Touching either shoulder blade with the hand, picking up a full glass of water, unbuttoning a button, and cutting with a knife. Improvement was defined as the ability to perform more such functions at discharge compared with admission.
Improvement in gait pattern | The day of discharge from hospitalization (average 10 days)
  Increase of one level on the Holden scale between admission and discharge
Residence change | The day of discharge from hospitalization (average 10 days)
  Institutionalisation and residence change because of a new disability

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Albacete, Spain

REFERENCES:
- [Result] Abizanda P, Navarro JL, Romero L, Leon M, Sanchez-Jurado PM, Dominguez L. Upper extremity function, an independent predictor of adverse events in hospitalized elderly. Gerontology. 2007;53(5):267-73. doi: 10.1159/000102541. Epub 2007 May 8. PMID 17495480